CLINICAL TRIAL: NCT06541509
Title: A Pilot Clinical Trial Investigating Underlying Mechanisms of Semaglutide Therapy in Heart Failure Patients
Brief Title: Mechanisms of Semaglutide Therapy in Heart Failure Patients
Acronym: SEMAHEART
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Stanford University (Other); Greenstone Biosciences (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEMAHEART
Record Dates: First submitted 2024-07-11; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure; Obesity
MeSH Terms: conditions — Heart Failure; Obesity | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Semaglutide Therapy (Experimental): Timepoints:
  * Baseline (Week 0)
  * Week 2 (Visit 1)
  * Week 4 (Visit 2)
  * Week 12 (Visit 3)
  * Week 16 (Visit 4)
  Medication Schedule:
  Subcutaneous semaglutide (Ozempyc, Novo Nordisk A/S Bagsvaerd, Denmark) First 2 weeks: Semaglutide; 0.25 mg weekly Second 2 weeks: Semaglutide; 0.5 mg weekly Remaining 12 weeks: Semaglutide; 1 mg weekly
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — 10 overweight patients with heart failure will be enrolled, including 5 patients with heart failure with preserved ejection fraction (HFpEF) and 5 patients with heart failure with reduced ejection fraction (HFrEF). The diagnosis of HFpEF and HFrEF will be based on the most recent European Society of Cardiology guidelines for the diagnosis and treatment of heart failure.
  After their baseline blood sample collections, all participants will receive once-weekly subcutaneous semaglutide (Ozempyc, Novo Nordisk A/S Bagsvaerd, Denmark) at a dose of 0.25 mg for 2 weeks, 0.5 mg for 2 weeks, and then 1.0 mg for a period of 12 weeks. At the end of the 3-month and 4-month period, blood sample collections will be repeated. All blood samples will be sent to Stanford Cardiovascular Institute for further analyses. At baseline, and again at 4 months transthoracic echocardiography, 6-minute walk test, and body composition assessment will be performed.

SUMMARY:
Semaglutide is a glucagon-like peptide-1 (GLP-1) receptor agonist, primarily used for treatment of type-2 diabetes mellitus. GLP-1 receptors are present on pancreatic islet β-cells, δ-cells and α-cells. Their stimulation increases insulin and somatostatin secretion, and decreases glucagon secretion. In addition, GLP-1 receptor agonists appear to have multiple extrapancreatic actions, which remain poorly defined. In large clinical trials, semaglutide improved the outcomes in obese patients, patients with heart failure with preserved ejection fraction, and decreased the heart failure hospitalizations in patients with type 2 diabetes. The aim of the present study is to investigate the underlying mechanisms of the beneficial clinical effects of semaglutide in the setting of chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-80 years
* Presence of heart failure
* Body-mass index 27 kg/m2 or greater
* Stable optimally tolerated dosages of heart failure therapies for 3 months
* N-terminal pro B-type natriuretic peptide levels >350 pg/mL

Exclusion Criteria:

* Presence of type 1 or type 2 diabetes or glycated haemoglobin higher than 6.5%
* Pregnancy or potential to become pregnant
* Cancer
* Liver dysfunction (aspartate aminotransferase and/or alanine aminotransferase > 3 times upper limits of normal or total bilirubin greater than 1.5 times upper limits of normal)
* Renal dysfunction (estimated glomerular filtration rate less than 25 mL/min/1.73 m2)
* Hospitalization in the past 3 months for reasons other than heart failure
* New York Heart Association (NYHA) functional class I or functional class IV symptoms.
* Prior or planned bariatric surgery
* Self-reported change in body weight >11 lbs (5 kg) within 3 months before enrollment
* Acute or chronic infection

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Interleukin-6 (IL-6) | 4 months
  Measured using enzyme linked immunosorbent assay (ELISA). Units of Measure: picograms per milliliter (pg/mL).
Interleukin-8 (IL-8) | 4 months
  Measured using ELISA. Units of Measure: picograms per milliliter (pg/mL).
Tumor Necrosis Factor-alpha (TNF-α) | 4 months
  Measured using ELISA. Units of Measure: picograms per milliliter (pg/mL).
Interferon-gamma (IFN-γ) | 4 months
  Measured using ELISA. Units of Measure: picograms per milliliter (pg/mL).
B-type Natriuretic Peptide (BNP) | 4 months
  Measured using immunoassay. Units of Measure: picograms per milliliter (pg/mL).
C-reactive Protein (CRP) | 4 months
  Measured using immunoassay. Units of Measure: picograms per milliliter (pg/mL).
Hemoglobin A1C (HgA1C) | 4 months
  Measured using standard laboratory methods. Units of Measure: percent (%).
Complete Blood Count (CBC) | 4 months
  Measured using automated hematology analyzer. CBC parameters will be measured in their respective units (e.g., cells per microliter).
Comprehensive Metabolic Panel (Chem 7) | 4 months
  Measured using standard laboratory methods. Chem 7 parameters will be measured in their respective units (e.g., mg/dL, U/L).
Liver Function Tests (LFT) | 4 months
  Measured using standard laboratory methods. LFT parameters will be measured in their respective units (e.g., mg/dL, U/L).
Body mass index | 4 months
  Patient weight will be measured in kilograms and height will be measured in meters. Body mass index (BMI) will be calculated according to the standard formula: weight in kilograms divided by height in meters squared.

SECONDARY OUTCOMES:
Left ventricular end-systolic volume (LVESV) | 4 months
  Measured using echocardiography. Units of measure: mililiter (mL)
Left ventricular end-diastolic volume (LVEDV) | 4 months
  Measured using echocardiography. Units of measure: mililiter (mL)
Myocardial mass | 4 months
  Measured using echocardiography. Units of measure: gram (g)
Left ventricular ejection fraction (LVEF) | 4 months
  Measured using echocardiography. Units of measure: percent (%)
Left ventricular filling pressures (E/e') | 4 months
  Measured using echocardiography. Units of measure: numerical value
Global longitudinal strain (GLS) | 4 months
  Measured using echocardiography. Units of measure: percent (%)
Exercise capacity | 4 months
  Measured by 6-minute walk test distance Units of measure: meter (m)
Lean body mass | 4 months
  Measured using dual-energy X-ray absorptiometry Units of measure: gram (g)
Fat mass | 4 months
  Measured using dual-energy X-ray absorptiometry Units of measure: gram (g)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Greenstone Biosciences, Palo Alto, California
  - Stanford Cardiovascular Institute, Stanford, California
- University Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No